CLINICAL TRIAL: NCT02154074
Title: Dexmedetomidine Influence on the Level of Perioperative Blood Glucose and Insulin of Elderly Diabetes Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dexmedetomidine 20140527
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Perioperative Blood Glucose and Insulin
Keywords: Dexmedetomidine perioperative blood glucose and insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Isoflurane; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- N1 group: Isoflurane & saline (Active Comparator): for normal patients: inhale Isoflurane + the same volume of saline during operation
  Interventions: Drug: general anesthesia induction; Drug: Isoflurane; Drug: normal saline
- N2 group: Isoflurane & Dexmedetomidine (Experimental): for normal patients: inhale Isoflurane + intravenous pumping Dexmedetomidine during operation
  Interventions: Drug: general anesthesia induction; Drug: Isoflurane; Drug: Dexmedetomidine
- D1 group: Isoflurane & saline (Active Comparator): for diabetes patients: inhale Isoflurane + the same volume of saline during operation
  Interventions: Drug: general anesthesia induction; Drug: Isoflurane; Drug: normal saline
- D2 group: Isoflurane & Dexmedetomidi (Experimental): for diabetes patients: inhale Isoflurane + intravenous pumping Dexmedetomidine during operation
  Interventions: Drug: general anesthesia induction; Drug: Isoflurane; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: general anesthesia induction — general anesthesia induction: midazolam 0.1mg/Kg, sufentanil 1ug/Kg, cisatracurium 0.15mg/Kg, and then immediatly administrate etomidate 0.2 mg/Kg
Drug: Isoflurane — inhale Isoflurane 1.5MAC
Drug: Dexmedetomidine — anesthesia induction period: intravenous pumping Dexmedetomidine 4ug/Kg/h; after 10 minutes,turn to 0.4ug/Kg/h.
  Arms: D2 group: Isoflurane & Dexmedetomidi; N2 group: Isoflurane & Dexmedetomidine
Drug: normal saline — the same volume of saline + Isoflurane during operation
  Arms: D1 group: Isoflurane & saline; N1 group: Isoflurane & saline

SUMMARY:
Dexmedetomidine is a kind of high selectivity alpha 2 agonists adrenaline, can inhibit the activity of sympathetic nerve, alleviate pain,and improve cardiovascular stability in the operation period. Dexmedetomidine have influence on perioperative stress response and immune function,but it is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 80 years old;
* Type 2 diabetes;
* Not use insulin treatment;
* Onging general anesthesia surgery;
* Surgery time 1-3 hours

Exclusion Criteria:

* ASA classification > class II;
* Hypertension;
* Serious central nervous system diseases (acute stroke, uncontrolled seizures, -Severe dementia);
* Unstable angina and acute myocardial infarction;
* Allergy to investigational drug;
* Hepatic and renal dysfunction

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
blood glucose | from the day before surgery to 24 hours after surgery
  measure blood glucose at 3 time points,the day before surgery,Intraoperative(1 hour after surgery begain),one day after surgery(24 hours after surgery); examine the concentration of blood glucose in serum.
level of blood insulin | from the day before surgery to 24 hours after surgery
  measure the level of blood insulin at 3 time points,the day before surgery,Intraoperative(1 hour after surgery begain),one day after surgery(24 hours after surgery); use ELISA to examine the concentration of blood insulin in serum.

SECONDARY OUTCOMES:
vital signs | duration of perioperative period
  measure the blood pressure(BP),heart rate(HR) and oxygen saturation(SpO2) in the perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- SecondXianJiaotongU, Xi’an, Shanxi, China